CLINICAL TRIAL: NCT01904474
Title: Internet Based Intervention Program for Obese Adolescents and Their Families(NEXT.STEP)
Brief Title: E-therapeutic Program for Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Santa Maria, Portugal (Other)
Collaborators: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Pedro Sousa, Dr., Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PTDC/DTP-PIC/0769/2012
Record Dates: First submitted 2013-07-09; First posted 2013-07-22 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Obesity
Keywords: obesity; overweight; technology; internet; intervention; adolescents
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Next.Step (Experimental): Experimental group participants, in addition to the standard treatment program are invited to get restricted access to the e-therapeutic platform (Next.Step), which includes a diverse set of resources, such as: educational resources (videos, brochures, menus, weekly tips, access to other links), self-monitoring (food, weight and physical activity records), social support (chats, discussion forums and personalized messages), interactive training modules (self-assessment quizzes, making their own diets) and motivational tools (personal goals planning, treatment progression registry, positive reinforcement).
  Intervention length will be 36 weeks (24 weeks of direct intervention with a follow-up of 12 weeks), being based on case management methodology.
  Interventions: Other: Next.Step - e-therapeutic intervention program
- Standard protocol (Active Comparator): The control group will follow the POC/HSM standard treatment protocol, which includes a baseline evaluation session with a paediatrician for initial screening, followed by appointments with the nutritionist and exercise physiologist. The second set of appointments will take place one month after for adjustments. After this, the adolescent will have appointments at 3, 6, 9 and 12 months. These adolescents will join a waiting list and nine months (36 weeks) after having started the standard treatment, they will receive the personal codes for accessing Next.Step.
  Interventions: Other: Standard treatment protocol

INTERVENTIONS:
Other: Next.Step - e-therapeutic intervention program
  Arms: Next.Step
Other: Standard treatment protocol
  Arms: Standard protocol

SUMMARY:
This study aims to:

I. Determine the e-therapeutic intervention program effectiveness compared with the standard treatment protocol, on both the behavioural change (treatment adherence and promotion of healthy lifestyles) and health impact (weight control and quality of life), based on a population of adolescents followed at Paediatric Obesity Clinic (POC) of Hospital de Santa Maria (HSM), Lisbon (Portugal).

II. Evaluate the health profile, treatment adherence, lifestyle and impact of weight on quality of life of this population.

III. Test the usability of an e-therapeutic platform for obese adolescents and their families.

DETAILED DESCRIPTION:
Information and Communications Technology (ICT) have been identified as important tools, allowing for health gains and reducing costs. They have been associated with positive results in terms of efficiency, effectiveness, equity, accessibility and quality of the provided care/services (Alcañiz et al., 2009; Baulch et al., 2008; Cottrell, 2005; Grohol, 1999). The existence of accurate, reliable, structured and relevant information, available when and where is needed, enables professionals and consumers to make informed and timely decisions (High Commissioner for Health, 2010; Organization for Economic Cooperation and Development, 2010).

This project was designed according to the national guidelines (Direção-Geral da Saúde, 2005), and has the potential to become a relevant educational and intervention instrument. Its content may be adapted to the needs and expectations of target groups. Strategies as problem solving reinforced by the e-therapeutic programme may enable participants to overcome barriers to adherence and thereby enhance treatment-induced weight losses (Murawski et al., 2009). Moreover, this project will allow to: a) Obtain relevant information about patients and their progress, enabling health professionals to interpret the inputs and send feedback in real time, b) Tailor therapeutic strategies to individual responses, c) Monitor individual progress.

This study is designed as a randomized clinical trial. The experimental group will follow the standard treatment protocol and, additionally, receive free access to the e-therapeutic platform (Next.Step) for 24 weeks. The control group participants will follow the standard treatment protocol and join a waiting list for entering the Next.Step.

Based on the literature review and on the contribution of the Nola Pender's Health Promotion reference model (Pender et al., 2010), investigators will look for empirical evidence for the general investigation hypothesis: treatment adherence, healthy lifestyles, quality of life and weight control of obese adolescents are positively influenced by this intervention program.

ELIGIBILITY:
Inclusion Criteria:

* patients from POC/HSM
* aged between 12 and 18 years
* BMI percentile ≥ 95th
* internet access at least once a week

Exclusion Criteria:

* presence of severe psychopathology
* inability to communicate in writing
* pregnancy
* having been proposed for bariatric surgery

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Body mass index percentile | 24 weeks
  Change in BMI percentile from baseline to 24 weeks. Height and weight will be used to calculate BMI percentile, adjusted for age and gender.

SECONDARY OUTCOMES:
Change in physical activity | 24 weeks
  Change in physical activity from baseline to 24 weeks, measure in self-reported hours/week
Change in sedentary lifestyle | 24 weeks
  Change in physical activity from baseline to 24 weeks, measure in self-reported hours/week of screen time
Change in body image | 24 weeks
  Change in body image silhouette perception from baseline to 24 weeks
Next.Step Usability | 24 weeks
  Perception of usability of the Next.Step platform measure with a self-reported instrument (NSUQ - Next.Step Usability Questionnaire)
Change in weight specific quality of life | 24 weeks
  Change in weight specific quality of life from baseline to 24 weeks, evaluated with a self-report instrument (IWQOL - Impact of Weight on Quality of Life)
Change in adherence to weight control | 24 weeks
  Change in adherence to weight control from baseline to 24 weeks, evaluated with a self-report instrument (AWCQ - Adherence to Weight Control Questionnaire)
Change in Lifestyle Profile | 24 weeks
  Change in Lifestyle Profile from baseline to 24 weeks, evaluated with a self-report instrument (ALP - Adolescent Lifestyle Profile).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Sousa, Msc, Study Chair — Instituto Politécnico de Leiria; Helena R Fonseca, PhD, Principal Investigator — Hospital de Santa Maria, Portugal; Pedro J Gaspar, PhD, Study Chair — Instituto Politécnico de Leiria
Locations (2):
- Portugal (2):
  - Instituto Politécnico de Leiria, Leiria
  - Hospital de Santa Maria, Lisbon

REFERENCES:
- [Background] Alcañiz M, Botella C, Baños R, Zaragoza I, Guixeres J. The Intelligent e-Therapy system: a new paradigm for telepsychology and cybertherapy. British Journal of Guidance & Counselling 37(3): 287-296, 2009.
- [Background] Baulch J, Chester A, Brennan L. Treatment Alternatives for Overweight and Obesity: The Role of Online Interventions. Behaviour Change 25(1): 1-14, 2008.
- [Background] Cottrell S. E-therapy: the future? Healthcare Counselling & Psychotherapy Journal 5(1): 18-21, 2005.
- [Background] Direção-Geral da Saúde. Programa Nacional de Combate à Obesidade. Circular Normativa nº 03/DGCG de 17/03/2005.
- [Background] Grohol JH. Best practices in e-therapy: Definition & Scope of e-therapy. 1999. Available at: www.psychcentral.com/best/best3.htm (accessed 12 Feb 2012).
- [Background] High Commissioner for Health [Alto Comissariado da Saúde]. Plano Nacional de Saúde 2011-2016: Tecnologias de Informação e Comunicação, 2010. Available at: www.acs.min-saude.pt/pns2011-2016/files/2010/07/TIC4.pdf (accessed 12 Fev 2012).
- [Background] Murawski ME, Milsom VA, Ross KM, Rickel KA, DeBraganza N, Gibbons LM, Perri MG. Problem solving, treatment adherence, and weight-loss outcome among women participating in lifestyle treatment for obesity. Eat Behav. 2009 Aug;10(3):146-51. doi: 10.1016/j.eatbeh.2009.03.005. Epub 2009 Mar 29. PMID 19665096
- [Background] Organization for Economic Cooperation and Development. Improving health sector efficiency - The role of information and communication technologies. Paris: OECD Health Policy Studie, 2010.
- [Background] Pender N, Murdaugh C, Parsons M. Health Promotion in Nursing Practice (6th ed.). Upper Saddle River, NJ: Pearson/Prentice-Hall.
- [Derived] Fonseca H, Prioste A, Sousa P, Gaspar P, Machado Mdo C. Effectiveness analysis of an internet-based intervention for overweight adolescents: next steps for researchers and clinicians. BMC Obes. 2016 Mar 9;3:15. doi: 10.1186/s40608-016-0094-4. eCollection 2016. PMID 26966545
- [Derived] Sousa P, Fonseca H, Gaspar P, Gaspar F. Controlled trial of an Internet-based intervention for overweight teens (Next.Step): effectiveness analysis. Eur J Pediatr. 2015 Sep;174(9):1143-57. doi: 10.1007/s00431-015-2502-z. Epub 2015 Mar 14. PMID 25772743